CLINICAL TRIAL: NCT06651671
Title: Measuring Muscle Tone in Thoracic Myofascial Release with the MyotonPRO Device
Brief Title: Tissue Changes Following Thoracic Myofascial Release
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rowan University (Other)
Responsible Party: Principal Investigator, Alexander King, DO, Program Director, Assistant Professor, Rowan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rowan-PRO-2022-348
Record Dates: First submitted 2024-09-27; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Myofascial Dysfunction; Myofascial Release
Keywords: Myofascial Release; Osteopathic Manipulative Medicine
MeSH Terms: interventions — Myofascial Release Therapy; salicylhydroxamic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment; MFR (Experimental): The treatment group received 30 seconds of direct and indirect myofascial release performed by the same practicing osteopathic physician.
  Interventions: Procedure: Myofascial release
- Control (Sham Comparator): The sham control group received one minute of light sham touch performed by a medical student.
  Interventions: Procedure: Sham (No Treatment)

INTERVENTIONS:
Procedure: Myofascial release — THe treatment group was instructed to lay prone on the treatment table such that the skin on their upper back was visible. Participants then received direct and indirect myofascial release for 30 seconds each, performed by the same osteopathic physician.
  Arms: Treatment; MFR
Procedure: Sham (No Treatment) — The medical student gently placed their hands on the patients back for 60 seconds without manipulating the tissue in any way.
  Arms: Control

SUMMARY:
Brief Summary:

The goal of this clinical trial is to determine the efficacy of myofascial release in altering the parameters of muscle tone, stiffness, and viscoelasticity in young adults. The main questions it aims to answer are:

What is the efficacy of myofascial release in altering muscle tone, stiffness, and viscoelasticity? What is the efficacy of light hands-on sham as a control? Are there differences in these parameters between men and women? What is the reliability of MyotonPro use in young adults? Researchers will randomly allocate and compare the treatment group, which receives osteopathic manipulative medicine (OMM) in the form of 30 seconds of indirect myofascial release followed by 30 seconds of direct myofascial release, to the control group, which receives 1 minute of light hands-on traps placebo, to see if there are differences in muscle tone, stiffness, and viscoelasticity.

DETAILED DESCRIPTION:
Objectives:

The primary objective was to determine the efficacy of myofascial release in altering the parameters of muscle tone, stiffness, and viscoelasticity. The secondary objectives are to determine the efficacy of light hands-on sham as a control, study the differences in parameters between men and women, and measure the reliability of MyotonPro use in young adults.

Eligibility Criteria:

Participants have to be aged 18 to 35 years old. Participants should not have current thoracic spine injuries such as compression fractures or prior thoracic spinal fusions.

Exclusion criteria included current or prior thoracic injury or surgery, as well as a BMI of less than 30.0. This exclusion was to maintain study validity, considering that >20mm of subcutaneous fat over the target muscle skews the data per the MyotonPro user manual.

Participants will be required to have a target muscle thickness >3mm, which was met as the trapezius was the target muscle for assessment.

Participants will report their height and weight during measurement, and if they did not meet the criteria, their data will be excluded without notification.

Study Design:

Before treatment, participants' trapezius muscle will be marked and measured at two inches lateral to the level of the T3 spinous process using a skin-safe marker. Muscle tone, stiffness, and viscoelasticity will be measured with the MyotonPRO in an average of five continuous measurements. Treatment and myotonometric assessment will be performed either shirtless or in a sports bra in the prone position with participants' arms by their side. Sterilization protocols will be followed between uses, and gowns will be available for participant comfort and privacy. Informed consent will be signed upon arrival, and five minutes will be given for consideration or questions.

Participants will be randomly and evenly separated into control (n = 30) and treatment (n = 30) groups by an online randomizer. The treatment group will receive both direct and indirect myofascial release for thirty seconds each, performed by the same practicing osteopathic physician. The control group will receive light sham touch for one minute performed by a medical student. The sham touch protocol has been shown to be an effective control method in prior studies.

Treatment Protocol:

Participants lay prone on the table. The operator stands at the dominant eye side of the table and palpated bilaterally over the thoracic spine, specifically two inches lateral to the level of T3, to assess the trapezius muscle.

This location will be marked for precise pre-post treatment testing and palpated for the preferred direction of myofascial tissues.

The technique involves placing tissue into its barriers of restriction for direct myofascial release or guiding myofascial into its preference for indirect release.

Tissues will be stacked into their direct bind for 30 seconds and then indirect bind for 30 seconds.

Post-Treatment Assessment:

Immediately following the treatment protocol, muscle tone, stiffness, and elasticity will be re-assessed using the MyotonPro. This device objectively quantifies muscle parameters by pressing a superficial probe onto the skin surface, producing a 0.6N force, and measuring the rate of probe acceleration and resistance. The device auto-corrects for human error and invalidates measurements if excessive movement is detected.

For reliability, the device will be operated by a single medical student experienced with its use. The phrase "stay as relaxed as possible" was used before each measurement, and each subject was assessed in the same prone position. Subjective symptom improvement data was not collected due to lack of power in this study.

Statistical Analysis and Measures:

A paired t-test will be conducted using the 2024 JASP computer statistical software (Version 0.19.0) to compare pre- and post-treatment muscle tone values within each group for the three variables. Sample size calculation was done using G*power V3.1. Normality assessment and Wilcoxon signed-rank test were used when necessary. Effect size was measured and reported with Cohen's D. Results were represented with bar plots to visualize changes in muscle tone, stiffness, and viscoelasticity.

Blinding:

Single blinding will be applied; participants will be unaware of their treatment group, though the study team will know. Both groups will receive baseline MyotonPro measurements, designed treatment, and post-treatment measurement. No follow-up or end-of-study visit will be required.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 year old healthy participants

Exclusion Criteria:

* BMI >30
* No current thoracic spine injuries such as compression fractures or spinal fusions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Tissue Biomechanical Parameters | Baseline will be assessed Immediately pre-treatment, with follow up assessed immediately after the intervention
  Myofascial Tone assessed using a Myotonometer
Tissue Biomechanical Parameters | Baseline will be assessed Immediately pre-treatment, with follow up assessed immediately after the intervention
  Myofascial Stiffness assessed using a Myotonometer
Tissue Biomechanical Parameters | Baseline will be assessed Immediately pre-treatment, with follow up assessed immediately after the intervention
  Myofascial Elasticity assessed using a Myotonometer

CONTACTS AND LOCATIONS:
Overall Officials: Alexander King, DO, Principal Investigator — Rowan-Virtua School of osteopathic medicine
Locations (1):
- Rowan University, Neuromuscular Institute, Stratford, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Data no longer retained for confidentiality purposes